CLINICAL TRIAL: NCT03824574
Title: Cephalometric Evaluation of a Clear Mandibular Advancement Appliance Based on the Twin-block Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa Zaky, Lecturer of Orthodontics, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AinShamsUOrthodontics
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Skeletal Malocclusion
Keywords: Functional appliance; skeletal class II; mandibular deficiency; twin-block; Growing patients; Clear appliance; Aligner
MeSH Terms: conditions — Micrognathism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Subjects receiving the clear mandibular advancement appliance
  Interventions: Device: Clear Mandibular Advancement Appliance

INTERVENTIONS:
Device: Clear Mandibular Advancement Appliance — Clear Mandibular Advancement Appliance for treatment of skeletal class II patients with retrognathic mandible

SUMMARY:
This study evaluates the cephalometric effects of a clear mandibular advancement appliance for the treatment of skeletal class II growing patients suffering from mandibular deficiency.

DETAILED DESCRIPTION:
A Clear mandibular advancement appliance is constructed comprised of a clear dental splint of 1.5 mm thickness adapted on the patient's teeth. This is followed by the construction of acrylic bite ramps bonded over the splints. The bite ramps are constructed as such when the patient bites into occlusion, he/she has to advance the mandible to bring the two parts of the appliance together. Lateral cephalometric radiographs were obtained pre and post-treatment to evaluate the effects on the patient's maxilla, mandible and dentition.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Female subjects.
2. Chronological age: All recruited subjects were between the ages of 8-12 years.
3. Anteroposterior skeletal relationship: Subjects with skeletal Class II malocclusion with normal maxilla and retrognathic mandible were selected. This was confirmed using lateral cephalometric radiographic analysis with the following parameters: decreased effective mandibular length (Co-Gn) according to McNamara composite , SNB<78, SNA=82+2.
4. Dental characteristics:

   * Angle Class II molar relationship ranging from edge to edge to full unit Class II.
   * Overjet ranging between 5-10 mm.
   * Absence of posterior crossbite and/or tendency for posterior crossbite.
5. Skeletal maturation stage: The growth stage for all subjects was selected to be before or at the prepubertal growth spurt. This was confirmed by cervical vertebral maturation analysis from the lateral cephalometric radiograph. The cervical vertebrae maturation stage required was Cervical Vertebrae Maturation stage 2-3 according to the cervical vertebrae maturation index by Baccetti et al. allowing sufficient time before the end of the growth spurt.
6. No previous history of orthodontic treatment.
7. Absence of systemic diseases affecting growth or craniofacial development. -

Exclusion Criteria:

-

Ages: 8 Years to 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-03-04 (Actual)

PRIMARY OUTCOMES:
Effective Mandibular Length | 12 months
  Condylion-Gnathion
Mandible to cranial base | 12 months
  Sella-Nasion-B point
Effective maxillary length | 12 months
  Condylion-A point
Maxilla to cranial base | 12 months
  Sella-Nasion-A point

SECONDARY OUTCOMES:
Lower incisor inclination | 12 months
  Lower incisor to mandibular plane
Lower incisor AP position | 12 months
  Lower incisor Anteroposterior position
Upper incisor inclination | 12 months
  Upper incisor to palatal plane
Upper incisor AP position | 12 months
  Upper incisor Anteroposterior position
Profile convexity | 12 months
  N'Sn/Sn-Pog'
Lip protrusion | 12 months
  Ls-E plane
Chin position | 12 months
  Soft tissue Pogonion position

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jena AK, Duggal R, Parkash H. Skeletal and dentoalveolar effects of Twin-block and bionator appliances in the treatment of Class II malocclusion: a comparative study. Am J Orthod Dentofacial Orthop. 2006 Nov;130(5):594-602. doi: 10.1016/j.ajodo.2005.02.025. PMID 17110256
- [Background] Teuscher U. A growth-related concept for skeletal class II treatment. Am J Orthod. 1978 Sep;74(3):258-75. doi: 10.1016/0002-9416(78)90202-6. PMID 281130
- [Background] Lv Y, Yan B, Wang L. Two-phase treatment of skeletal class II malocclusion with the combination of the twin-block appliance and high-pull headgear. Am J Orthod Dentofacial Orthop. 2012 Aug;142(2):246-55. doi: 10.1016/j.ajodo.2010.12.024. PMID 22858335
- [Background] O'Brien K, Macfarlane T, Wright J, Conboy F, Appelbe P, Birnie D, Chadwick S, Connolly I, Hammond M, Harradine N, Lewis D, Littlewood S, McDade C, Mitchell L, Murray A, O'Neill J, Sandler J, Read M, Robinson S, Shaw I, Turbill E. Early treatment for Class II malocclusion and perceived improvements in facial profile. Am J Orthod Dentofacial Orthop. 2009 May;135(5):580-5. doi: 10.1016/j.ajodo.2008.02.020. PMID 19409340
- [Background] Tulloch JF, Phillips C, Koch G, Proffit WR. The effect of early intervention on skeletal pattern in Class II malocclusion: a randomized clinical trial. Am J Orthod Dentofacial Orthop. 1997 Apr;111(4):391-400. doi: 10.1016/s0889-5406(97)80021-2. PMID 9109584
- [Background] Cozza P, Baccetti T, Franchi L, De Toffol L, McNamara JA Jr. Mandibular changes produced by functional appliances in Class II malocclusion: a systematic review. Am J Orthod Dentofacial Orthop. 2006 May;129(5):599.e1-12; discussion e1-6. doi: 10.1016/j.ajodo.2005.11.010. PMID 16679196
- [Background] Baccetti T, Franchi L, Toth LR, McNamara JA Jr. Treatment timing for Twin-block therapy. Am J Orthod Dentofacial Orthop. 2000 Aug;118(2):159-70. doi: 10.1067/mod.2000.105571. PMID 10935956
- [Background] Clark WJ. The twin block technique. A functional orthopedic appliance system. Am J Orthod Dentofacial Orthop. 1988 Jan;93(1):1-18. doi: 10.1016/0889-5406(88)90188-6. No abstract available. PMID 3422118
- [Background] Toth LR, McNamara JA Jr. Treatment effects produced by the twin-block appliance and the FR-2 appliance of Frankel compared with an untreated Class II sample. Am J Orthod Dentofacial Orthop. 1999 Dec;116(6):597-609. doi: 10.1016/s0889-5406(99)70193-9. PMID 10587592
- [Background] Trenouth MJ. Cephalometric evaluation of the Twin-block appliance in the treatment of Class II Division 1 malocclusion with matched normative growth data. Am J Orthod Dentofacial Orthop. 2000 Jan;117(1):54-9. doi: 10.1016/s0889-5406(00)70248-4. PMID 10629520
- [Background] Mills CM, McCulloch KJ. Posttreatment changes after successful correction of Class II malocclusions with the twin block appliance. Am J Orthod Dentofacial Orthop. 2000 Jul;118(1):24-33. doi: 10.1067/mod.2000.104902. PMID 10893470
- [Background] Singh GD, Hodge MR. Bimaxillary morphometry of patients with class II division 1 malocclusion treated with twin block appliances. Angle Orthod. 2002 Oct;72(5):402-9. doi: 10.1043/0003-3219(2002)0722.0.CO;2. PMID 12401048
- [Background] Schaefer AT, McNamara JA Jr, Franchi L, Baccetti T. A cephalometric comparison of treatment with the Twin-block and stainless steel crown Herbst appliances followed by fixed appliance therapy. Am J Orthod Dentofacial Orthop. 2004 Jul;126(1):7-15. doi: 10.1016/j.ajodo.2003.06.017. PMID 15224053
- [Background] O'Brien K, Wright J, Conboy F, Sanjie Y, Mandall N, Chadwick S, Connolly I, Cook P, Birnie D, Hammond M, Harradine N, Lewis D, McDade C, Mitchell L, Murray A, O'Neill J, Read M, Robinson S, Roberts-Harry D, Sandler J, Shaw I. Effectiveness of treatment for Class II malocclusion with the Herbst or twin-block appliances: a randomized, controlled trial. Am J Orthod Dentofacial Orthop. 2003 Aug;124(2):128-37. doi: 10.1016/s0889-5406(03)00345-7. PMID 12923506
- [Background] Flores-Mir C, Major PW. Cephalometric facial soft tissue changes with the twin block appliance in Class II division 1 malocclusion patients. A systematic review. Angle Orthod. 2006 Sep;76(5):876-81. doi: 10.1043/0003-3219(2006)076[0876:CFSTCW]2.0.CO;2. PMID 17029526
- [Background] Khoja A, Fida M, Shaikh A. Cephalometric evaluation of the effects of the Twin Block appliance in subjects with Class II, Division 1 malocclusion amongst different cervical vertebral maturation stages. Dental Press J Orthod. 2016 Jun;21(3):73-84. doi: 10.1590/2177-6709.21.3.073-084.oar. PMID 27409656
- [Background] Mills CM, McCulloch KJ. Treatment effects of the twin block appliance: a cephalometric study. Am J Orthod Dentofacial Orthop. 1998 Jul;114(1):15-24. doi: 10.1016/s0889-5406(98)70232-x. PMID 9674675